CLINICAL TRIAL: NCT02409225
Title: Remote Supervision to Decrease Hospitalization Rate (RESULT)
Brief Title: Remote Supervision to Decrease Hospitalization Rate
Acronym: RESULT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Silesian Centre for Heart Diseases (Other)
Collaborators: National Center for Research and Development, Poland (Other)
Responsible Party: Principal Investigator, Lech Polonski, Professor, PhD, MD, Silesian Centre for Heart Diseases
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STRATEGMED1\233221\3\NCBR\2014
Record Dates: First submitted 2015-03-26; First posted 2015-04-06 (Estimated); Last update posted 2017-07-25 (Actual); Status verified 2017-07

CONDITIONS: Heart Failure
Keywords: remote monitoring; ICD; CRT-D
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Home Monitoring (Experimental): Remote monitoring od ICD/CRT-D function and patient condition. Device: HM provided by St Jude Medical, Biotronik or Medtronic.
  Interventions: Device: Home Monitoring
- HM option not active. (Active Comparator): Regular visits in outpatient clinic. Device: no HM
  Interventions: Device: no Home Monitoring

INTERVENTIONS:
Device: Home Monitoring — Remote monitoring of ICD/CRT-D function and patient condition allow decreasing costs of treatment of patients with ICD/CRT-D (hospitalization, visits in outpatient clinic) and reducing waiting time for medical intervention (remote or in outpatient clinic).
  Arms: Home Monitoring
Device: no Home Monitoring — Patients with ICD/CRT-D devices provided by St Jude Medical, Biotronik or Medtronic with HM option switched off.
  Arms: HM option not active.

SUMMARY:
Purpose: Home monitoring (HM) services supplied by different manufacturers (St Jude Medical, Biotronik, Medtronic) enables trained medical staff (doctors, electrophysiology nurses and technicians) to safely follow-up patients with implanted ICD/CRT-D remotely, with omitting unnecessary visits in outpatient clinic, shortening time to medical intervention and therefore help to decrease hospitalization rate among those patients.

The RESULT study primary endpoint of the trial will be a composite of all-cause death or hospitalization due to cardiovascular reasons.

The primary technical endpoint is to construct and evaluate a unified and integrated platform for data collected from RM devices manufactured by different companies: Carelink™ (Medtronic®, Minneapolis, MN, USA), Merlin™ (Saint Jude Medical®, St. Paul, MN, USA) and Home Monitoring™ (Biotronik®, Berlin, Germany).

DETAILED DESCRIPTION:
The RESULT trial is a prospective, single-center, randomized, open label, parallel study. All consecutive patients with symptomatic HF and reduced ejection fraction (≤ 35%) with ICDs or CRT-Ds implanted accordingly to current ESC practice guidelines will be prospectively randomized in a 1:1 fashion to either a traditional or an RM-based follow-up model. Six hundred patients will be enrolled. The inclusion and exclusion criteria are shown in Table 1. The clinical status of patients will be estimated using the composite endpoint of all-cause death and hospitalization due to cardiovascular reasons. The study protocol has been approved by a local ethics committee and complies with the Declaration of Helsinki. A written informed consent will be obtained from all study participants. Primary endpoint The primary endpoint of the trial will be a composite of all-cause death or hospitalization due to cardiovascular reasons. Hospitalization for cardiovascular reasons should consist of:

* Hospitalization due to progression of heart failure.
* Hospitalization due to persistent arrhythmia (AF, VT).
* Hospitalization due to embolic episode.
* Hospitalization due to acute coronary syndrome. Every patient will be followed for at least 12 months after randomization. Assessment of hospitalization events for cardiovascular reasons will be performed according to a recently published consensus [13]. The final classification of hospital admissions due to cardiovascular reasons will be made by a blinded endpoints committee. The primary technical endpoint is to construct and evaluate a unified and integrated platform for data collected from RM devices manufactured by different companies: Carelink™ (Medtronic®, Minneapolis, MN, USA), Merlin™ (Saint Jude Medical®, St. Paul, MN, USA) and Home Monitoring™ (Biotronik®, Berlin, Germany). Secondary endpoints Both elements combined in the primary endpoint will be analyzed separately to estimate their relative impact on the primary endpoint.

The secondary endpoints include the following:

* All-cause death.
* Hospitalization due to cardiovascular reasons.
* Time to medical intervention in case of relevant incidents (arrhythmic, device malfunction, signs of HF decompensation).
* Average number of visits to an outpatient clinic (scheduled and unscheduled) per patient.
* Time to first unscheduled visit in an outpatient clinic.
* Incidence of inappropriate ICD shocks.
* Proportion of visits to outpatient clinics with relevant findings (necessity of changes of device programming or pharmacological therapy, rehospitalization, interventions, invasive procedures).
* Assessment of quality of life of living study participants according to the Minnesota Quality of Life Questionnaire.
* Cost-effectiveness, defined as the cost of hospitalizations and/or scheduled and unscheduled visits in both groups.

All consecutive patients after implantation of an ICD or CRT-D manufactured by St.

Jude Medical, Biotronik or Medtronic will undergo an initial evaluation. Patients who have given informed consent and who fulfill the inclusion/exclusion criteria will be screened. Randomization to the RM or control group will be conducted within 30 days after ICD or CRT-D implantation and after the final programming of sensing and stimulation parameters. The time of observation in both groups will be 12 months after randomization. In the RM group only, one follow-up visit will be planned 12 months after being enrolled in the trial. In the control group, follow-up visits will be planned at 3, 6, 9 and 12 months after being enrolled in the trial, according to the normal procedure in our center. Unscheduled visits in both groups can be initiated either by the patient or by the supervising staff. The limits of therapeutic intervention will be individualized depending on the clinical situation according to valid ESC guidelines and will include the following: modification of device settings, modification of pharmacotherapy and performing necessary invasive diagnostic and therapeutic procedures.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-80 years
2. EF≤35% prior to implantation
3. Period up to 30 days after implantation (ICD/CRT-D) according to ESC guidelines
4. Agreement for telemetric supervision
5. Informed consent for clinical trial.

Exclusion Criteria:

1. Existence of factors that may cause risk for lack of cooperation in trial regimen (distant residence, mental illness, lack of skills in operating simple electronic devices).
2. unavailability of mobile network service in the place of residence/stay.
3. Device implanted during intravenous administration of inotropic agents.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Actual)
Dates: Start 2014-09; Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
The primary endpoint of the trial will be composite: death for any reason or hospitalization due to cardiovascular reasons. | 12 months

SECONDARY OUTCOMES:
time to medical intervention in case of relevant incidents (arrhythmic, device malfunction, signs heart failure decompensation) in both arms of the study | 12 months
average number of visits in outpatient clinic (scheduled and unscheduled) per patient | 12 months
time to first unscheduled visit in outpatient clinic | 12 months
incidence of inappropriate ICD shocks | 12 months
proportion of visits in outpatient clinic with relevant findings (necessity of changes of device programming or pharmacological therapy, re-hospitalization, interventions, invasive procedures) | 12 months
changes in quality of life (Minnesota Quality of Life Questionnaire ) | baseline and after 12 months
costs of treatment of patients with implanted ICD/CRT-D in both arms of the study (hospitalization, control visits) | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Lech Polonski, PhD, MD, Principal Investigator — Silesian Centre for Heart Diseases
Locations (1):
- Silesian Centre for Heart Diseases, Zabrze, Silesian Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Tajstra M, Sokal A, Gadula-Gacek E, Kurek A, Wozniak A, Niedziela J, Adamowicz-Czoch E, Rozentryt P, Milewski K, Jachec W, Kalarus Z, Polonski L, Gasior M. Remote Supervision to Decrease Hospitalization Rate (RESULT) study in patients with implanted cardioverter-defibrillator. Europace. 2020 May 1;22(5):769-776. doi: 10.1093/europace/euaa072. PMID 32304216
- [Derived] Tajstra M, Sokal A, Gwozdz A, Wilczek M, Gacek A, Wojciechowski K, Gadula-Gacek E, Adamowicz-Czoch E, Chlosta-Niepieklo K, Milewski K, Rozentryt P, Kalarus Z, Gasior M, Polonski L. REmote SUpervision to Decrease HospitaLization RaTe. Unified and integrated platform for data collected from devices manufactured by different companies: Design and rationale of the RESULT study. Ann Noninvasive Electrocardiol. 2017 Jul;22(4):e12418. doi: 10.1111/anec.12418. Epub 2016 Dec 25. PMID 28019051